CLINICAL TRIAL: NCT03848403
Title: A Randomized Study to Investigate Injection-Site Pain Following Subcutaneous Injections of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation Using a Pre-filled Syringe in Healthy Subjects
Brief Title: Study of Ixekizumab in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: At the protocol-specified interim analysis, the sponsor decided to stop the trial.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 17139; I1F-MC-RHCS (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2020-07-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ixekizumab (Reference) (Experimental): Reference formulation 80 milligram (mg) ixekizumab administered as a subcutaneous (SC) injection in a prefilled syringe in one of three study periods.
  Interventions: Biological: Ixekizumab
- Ixekizumab (Test 1) (Experimental): Test 1 formulation 80 mg ixekizumab administered as an SC injection in a prefilled syringe in one of three study periods.
  Interventions: Biological: Ixekizumab
- Ixekizumab (Test 2) (Experimental): Test 2 formulation 80 mg ixekizumab administered as an SC injection in a prefilled syringe in one of three study periods.
  Interventions: Biological: Ixekizumab

INTERVENTIONS:
Biological: Ixekizumab — Administered SC
  Other Names: LY2439821

SUMMARY:
The purpose of this study is to compare the tolerability of injections of each of 3 formulations of ixekizumab using a prefilled syringe. Information about any side effects (including injection site reactions [ISRs]) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants or female participants who agree not to get pregnant
* Are male participants or female participants with chronic, stable medical problems that, in the investigator's opinion, will not place the participant at increased risk by participating in the study

Exclusion Criteria:

* Have a significant history of, or current, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or hematologic disorders that in the opinion of the investigator poses an unacceptable risk to the participant if participating in the study
* Are allergic or hypersensitive to the study medicine
* Have dullness or loss of sensitivity on either side of your abdomen
* Have any condition that could affect pain perception from an injection
* Had a vaccination with a live vaccine within 12 months prior to the first check-in or intend to get a vaccine for tuberculosis within 12 months of completing treatment on this study
* Have any type of hepatitis, human immunodeficiency virus (HIV) infection, or other serious infection
* Show evidence of active or latent tuberculosis (TB)
* Presence of significant neuropsychiatric disorder or a recent history of depression
* Have excessive tattoos or scars over the abdomen or other factors such as rash or excessive folds of skin that would interfere with injection site assessments
* Have had any active or recent infection within 4 weeks of Day 1 that, in the opinion of the investigator would pose an unacceptable risk to the participant if participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance, Dallas, Texas
  - Covance Clinical Research Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chabra S, Gill BJ, Gallo G, Zhu D, Pitou C, Payne CD, Accioly A, Puig L. Ixekizumab Citrate-Free Formulation: Results from Two Clinical Trials. Adv Ther. 2022 Jun;39(6):2862-2872. doi: 10.1007/s12325-022-02126-0. Epub 2022 Apr 21. PMID 35449322

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to a treatment sequence in one of three periods. The study was stopped for some participants per sponsor decision and these participants did not move on to subsequent periods in the study at the protocol interim analysis.
Groups:
- Sequence 1: ABC: A: Reference formulation 80 milligram (mg) of Ixekizumab administered as a subcutaneous (SC) injection in a prefilled syringe in Period 1.
  B: Test 1 formulation 80 mg of Ixekizumab administered as an subcutaneous SC injection in a prefilled syringe in Period 2.
  C: Test 2 formulation 80 mg of Ixekizumab administered as an SC injection in a prefilled syringe in Period 3.
  Sequence 1: ABC (Reference, Test 1, then Test 2)
- Sequence 2: BCA: B: Test 1 formulation 80 mg of Ixekizumab administered as an SC injection in a prefilled syringe in Period 1.
  C: Test 2 formulation 80 mg of Ixekizumab administered as a SC injection in a prefilled syringe in Period 2.
  A: Reference formulation 80 mg of Ixekizumab administered as a SC injection in a prefilled syringe in Period 3.
  Sequence 2: BCA (Test 1, Test 2, Then Reference)
- Sequence 3: CAB: C: Test 2 formulation 80 mg of Ixekizumab administered as an SC injection in a prefilled syringe in Period 1.
  A: Reference: formulation 80 mg of Ixekizumab administered as a SC injection in a prefilled syringe in Period 2.
  B: Test 1 formulation 80 mg of Ixekizumab administered as an SC injection in a prefilled syringe in Period 3.
  Sequence 3: CAB (Test 2, Reference, Then Test 1)
Period: Period 1 (Day 1)
Arm/Group | Sequence 1: ABC | Sequence 2: BCA | Sequence 3: CAB
Started | 24 | 24 | 22
Received Intervention | 24 | 24 | 22
Completed | 24 | 24 | 22
Not Completed | 0 | 0 | 0
Period: Period 2 (Day 8)
Arm/Group | Sequence 1: ABC | Sequence 2: BCA | Sequence 3: CAB
Started | 24 | 24 | 22
Received at Least One Dose of Study Drug | 24 | 24 | 22
Completed | 15 | 15 | 15
Not Completed | 9 | 9 | 7
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Sponsor Decision | 8 | 6 | 5
Period: Period 3 (Day 15)
Arm/Group | Sequence 1: ABC | Sequence 2: BCA | Sequence 3: CAB
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of intervention.
Groups:
- All Study Participants: All randomized participants who received at least one 80 milligram (mg) dose of ixekizumab administered as an SC injection in a prefilled syringe in one of three periods.
Arm/Group | All Study Participants
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 41
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Injection Pain Visual Analog Scale (VAS) Score
Description: The injection pain VAS score is a participant administered single item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. The severity of pain was categorized by VAS pain score as: no pain (0), mild pain ≤ 30, moderate pain (>30 and ≤70), and severe pain (>70). Overall severity of participant's pain is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (worst imaginable pain).
Time Frame: Day 1, 8, and 15: Immediately (within 1 minute) after injection
Population: All randomized participants who received at least one dose of study drug in a treatment sequence.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Groups:
- Ixekizumab (Reference): Reference formulation ixekizumab 80 mg administered as a subcutaneous (SC) injection in a prefilled syringe in one of three study periods.
- Ixekizumab (Test 1): Test 1 formulation ixekizumab 80 mg administered as an SC injection in a prefilled syringe in one of three study periods.
- Ixekizumab (Test 2): Test 2 formulation ixekizumab administered as an SC injection in a prefilled syringe in one of three study periods.
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2)
Number analyzed (Participants) | 61 | 63 | 61
millimeter (mm) | 25.3 (24.7) | 3.3 (7.0) | 4.1 (8.2)
Statistical Analysis 1: Comparison: Ixekizumab (Reference) vs Ixekizumab (Test 1); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least Squares (LS) Means Difference = -21.69, 95% CI 2-sided [-26.90 to -16.48]
Statistical Analysis 2: Comparison: Ixekizumab (Reference) vs Ixekizumab (Test 2); Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Means Difference = -21.14, 95% CI 2-sided [-26.39 to -15.88]
Statistical Analysis 3: Comparison: Ixekizumab (Test 1) vs Ixekizumab (Test 2); Test type: Superiority; p = 0.8341, Mixed Models Analysis; LS Means Difference = 0.55, 95% CI 2-sided [-4.65 to 5.75]

ADVERSE EVENTS:
Time Frame: Up to 85 Days
Description: All randomized participants who received at least one dose of intervention.
Groups:
- Ixekizumab (Reference): Reference formulation 80 mg ixekizumab administered as a subcutaneous (SC) injection in a prefilled syringe in one of three study periods.
- Ixekizumab (Test 1): Test 1 formulation ixekizumab 80mg administered as an SC injection in a prefilled syringe in one of three study periods.
- Ixekizumab (Test 2): Test 2 formulation ixekizumab 80 mg administered as an SC injection in a prefilled syringe in one of three study periods.
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2)
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/63 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/63 | 0/61
Other Adverse Events (participants affected / at risk) | 3/61 | 5/63 | 6/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (Reference) (N=61) | Ixekizumab (Test 1) (N=63) | Ixekizumab (Test 2) (N=61)
Injection site reaction (General disorders) | 3 (3) | 5 (7) | 6 (8)

LIMITATIONS AND CAVEATS:
At protocol-specified interim analysis, the sponsor decided to stop trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03848403/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03848403/SAP_001.pdf